CLINICAL TRIAL: NCT00213980
Title: Bone Mineral Density Effects of Zoledronate in Postmenopausal Women With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CO99103; A534260 (Other: UW Madison); SMPH/MEDICINE/MEDICINE*H (Other: UW Madison)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2018-01-05 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer
Keywords: bone mineral density; postmenopausal women
MeSH Terms: conditions — Breast Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Observation (No Intervention): Observation only for 12 months
- Zoledronate (Active Comparator): Zoledronate
  Interventions: Drug: Zoledronate

INTERVENTIONS:
Drug: Zoledronate — 4 mg IV over 15 minutes administered once every 12 weeks times 4
  Other Names: Zometa
  Arms: Zoledronate

SUMMARY:
This is a two arm, double-blind randomized study looking at the effect of zoledronate, a bisphosphonate, on the bone mineral density (BMD) of postmenopausal women with breast cancer.

DETAILED DESCRIPTION:
This is a two arm, double-blind randomized study looking at the effect of zoledronate, a bisphosphonate, on the bone mineral density (BMD) of postmenopausal women with breast cancer. An approved bisphosphonate, alendronate, is of benefit in patients with osteoporosis, however, this agent has a roughly 30% incidence of gastrointestinal symptoms and up to 50% of patients may take the drug improperly, compromising absorption and potentially efficacy. Zoledronate is a heterocyclic imidazole third generation bisphosphonate, which is administered intravenously (IV) and has little toxicity. Zoledronate is more potent than alendronate, and because of its route of administration it does not have the problems of poor oral bioavailability and non-compliance.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women, Stage III or axillary node positive
* Currently disease free of breast cancer and other invasive malignancies at the time of registration
* No concurrent use of bisphosphonates

Exclusion Criteria:

* Metastatic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2000-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Mulkerin, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The University of Wisconsin Comprehensive Cancer Center (UWCCC) conducted a clinical trial of adjuvant ZA in postmenopausal women with high-risk breast cancer, open through the Wisconsin Oncology Network (WON). Participants were recruited from 2000 through 2007.
Groups:
- Zoledronic Acid (ZA): ZA
  Zoledronic acid (ZA): 4 mg IV over 15 minutes administered once every 12 weeks for 4 cycles
Period: Overall Study
Arm/Group | Observation | Zoledronic Acid (ZA)
Started | 32 | 36
Completed | 26 | 29
Not Completed | 6 | 7
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Disease progression | 0 | 2
Not completed — Developed ovarian cancer | 1 | 0
Not completed — Failed to obtain all 3 DXAs | 1 | 3

BASELINE CHARACTERISTICS:
Population: Postmenopausal women with stage II/III breast cancer diagnosed up to 5 years previous.
Groups:
- Total: Total of all reporting groups
Arm/Group | Observation | Zoledronic Acid (ZA) | Total
Number analyzed (Participants) | 32 | 36 | 68
Age, Continuous [Median (Full Range); unit: years] | 50.5 [37 to 65] | 54.5 [41 to 83] | 52.5 [37 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 36 | 68
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 32 | 35 | 67
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 36 | 68
Tumor Size [Count of Participants; unit: Participants]
  =< 2cm | 2 | 14 | 16
  2.1cm - 5cm | 18 | 11 | 29
  > 5cm | 9 | 9 | 18
  Inflammatory | 3 | 1 | 4
  Unknown | 0 | 1 | 1
Lymph Node Status [Count of Participants; unit: Participants]
  Node negative | 1 | 1 | 2
  Node positive | 31 | 35 | 66
Endocrine Therapy During Year 1 on Study [Count of Participants; unit: Participants]
  None | 3 | 5 | 8
  Tamoxifen or other SERM | 18 | 23 | 41
  Aromatase Inhibitor (AI) | 5 | 4 | 9
  Tamoxifen switched to AI during study year | 2 | 1 | 3
  No data available | 4 | 3 | 7
Performance Status [Count of Participants; unit: Participants] — Participants were required to have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2. ECOG performance is used to assess how a participant's disease is progressing, assess how the disease affects daily living abilities, and determine appropriate treatment and prognosis. A score of 0 is "fully active, able to carry on all pre-disease performance without restriction," and 2 is "ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours."
  Participants
    0 | 28 | 31 | 59
    1 | 3 | 4 | 7
    Unknown | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Bone Mineral Density (BMD) From Baseline to 1 Year
Description: To determine whether zoledronate 4 mg IV every 12 weeks x 4 doses is associated with increases in bone mineral density at the lumbar spine and femoral head, calculated from baseline and 1 year data. Participants who missed one or more DXA were not evaluated.
Time Frame: Up to 1 year
Population: Fifty-six participants (ZA = 29, Observation = 27) were evaluable based on completing DXAs at 0, 6, and 12 months.
Measure: Mean (95% Confidence Interval); unit: grams per cubic centimeter
Arm/Group | Zoledronic Acid (ZA) | Observation
Number analyzed (Participants) | 29 | 27
grams per cubic centimeter
  Lumbar Spine L1-L4 (L1-L4) | 0.048 [0.034 to 0.062] | 0.007 [-0.020 to 0.034]
  Femoral neck (FN) | 0.014 [0.002 to 0.027] | 0.005 [-0.012 to 0.023]
  Total femur (TF) | 0.019 [0.011 to 0.026] | 0.004 [-0.006 to 0.015]
  Trochanter (T) | 0.023 [0.013 to 0.34] | 0.005 [-0.007 to 0.017]
  Calcaneal (OC) | 0.010 [0.004 to 0.015] | 0.001 [-0.007 to 0.005]

2. Secondary Outcome: Rates of Metastases
Description: Determine whether zoledronate is associated in rates of bone, visceral, and all distant metastases.
Time Frame: Up to 1 year
Population: Data for this outcome measure was not collected.
Arm/Group | Zoledronic Acid (ZA) | Observation
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Survival
Description: Number of participants who survived from the start of treatment through off treatment, up to 10 years.
Time Frame: Up to 10 years
Population: Only participants who completed the trial (ZA = 29 and Observation = 26) were analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Zoledronic Acid (ZA) | Observation
Number analyzed (Participants) | 29 | 26
Participants | 24 | 22

4. Secondary Outcome: Clinical Toxicity of ZA
Description: Tolerability and side effects of ZA, measured by the number of participants experiencing adverse events.
Time Frame: Up to 1 year
Population: Data was collected for the ZA arm at 9 time points, and for the Observation arm at 2 time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Zoledronic Acid (ZA) | Observation
Number analyzed (Participants) | 36 | 32
Participants | 36 | 23

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for up to 48 weeks.
Description: Toxicity evaluation including telephone assessment occurred at 1 week after the start of each cycle.
  Toxicities for the Zoledronate arm were assessed at 9 time points, and toxicities for the Observation arm were assessed at 2 time points.
Arm/Group | Observation | Zoledronic Acid (ZA)
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/36
Other Adverse Events (participants affected / at risk) | 23/32 | 36/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observation (N=32) | Zoledronic Acid (ZA) (N=36)
Arthralgia (General disorders) | 3 (3) | 15 (30)
Back pain (General disorders) | 0 | 2 (3)
Bone pain (General disorders) | 0 | 5 (6)
Chest pain (Cardiac disorders) | 0 | 2 (2)
Constipation (Gastrointestinal disorders) | 0 | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 | 2 (3)
Edema (Cardiac disorders) | 2 (2) | 7 (11)
Eye pain (Eye disorders) | 0 | 2 (2)
Fatigue (General disorders) | 4 (4) | 27 (70)
Fever (General disorders) | 0 | 4 (4)
Headache (General disorders) | 0 | 20 (26)
Hot Flash (Endocrine disorders) | 13 (15) | 20 (36)
Lightheaded (Nervous system disorders) | 0 | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 28 (54)
Nausea (Gastrointestinal disorders) | 0 | 12 (15)
Neuropathy-sensory (Nervous system disorders) | 0 | 5 (11)
Pain (General disorders) | 4 (5) | 4 (6)
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 (3)
Rigors (General disorders) | 0 | 7 (9)
Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2 (2)
Vertigo (Nervous system disorders) | 0 | 4 (4)
Weight Gain (Investigations) | 0 | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No